CLINICAL TRIAL: NCT02725242
Title: A 12-week, Randomized, Parallel-group, Phase III Study Comparing the Efficacy of Once-daily Budesonide/Formoterol Turbuhaler (160/4.5 μg/d) and Twice-daily Budesonide Giona Easyhaler (400 μg/d) During Step-down Period in Well Controlled Asthma
Brief Title: Efficacy of Once-daily Budesonide/Formoterol Turbuhaler 4.5/160 µg in Step Down Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hat Yai Medical Education Center (Other)
Responsible Party: Principal Investigator, Narongwit Nakwan, Head of Pulmonology, Hat Yai Medical Education Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 064/2014
Record Dates: First submitted 2016-01-20; First posted 2016-03-31 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide; Formoterol Fumarate; Budesonide, Formoterol Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Once-daily budesonide/formoterol (160/4.5 μg/d) (Experimental): once-daily budesonide/formoterol (160/4.5 μg/d)
  Interventions: Drug: Budesonide/formoterol (160/4.5 μg/d)
- Twice-daily Budesonide (200μg) (Active Comparator): twice-daily Budesonide (400μg/d)
  Interventions: Drug: Budesonide (400μg/d)

INTERVENTIONS:
Drug: Budesonide/formoterol (160/4.5 μg/d) — After the patients who have all criteria, they will be randomization to take Budesonide/formoterol (160/4.5 μg/d)
  Other Names: Symbicort Turbuhaler (160/4.5 μg/d)
  Arms: Once-daily budesonide/formoterol (160/4.5 μg/d)
Drug: Budesonide (400μg/d) — After the patients who have all criteria, they will be randomization to take Budesonide (200 ug) twice daily
  Other Names: Giona Easyhaler
  Arms: Twice-daily Budesonide (200μg)

SUMMARY:
This study will evaluate the efficacy of Once-daily Budesonide/formoterol Turbuhaler 160/4.5 µg/d in the period of step down in well controlled asthmatic patient.

DETAILED DESCRIPTION:
The study will measure the efficacy of once daily low dose ICS/ LABA in well controlled asthmatic patient comparing with low dose ICS in step down circumstance.

ELIGIBILITY:
Inclusion Criteria:

* Asthmatic patients who have well controlled asthma at least 12 weeks with using budesonide/formoterol (160/4.5 μg/d) twice daily
* Age more than 18 year-old
* Patients who able to do spirometry without contraindication
* History smoking less than 10 pack-years

Exclusion Criteria:

* History of using systemic steroid previous 4 week and respiratory infection
* History of pulmonary tuberculosis with residual lung lesion by chest radiograph
* recent serious medical condition such as myocardial infarction, stroke, pneumonia etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2016-03; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Asthma Control Questionnaire (ACQ) score | Baseline and week 12
  Asthma Control Questionnaire (ACQ) that is 6 items of self-administered and 1 item of FEV1%. It has 7-point scale (=no impairment, 6= maximum impairment for symptoms and rescue use; and 7 categories for FEV1%). Scores range between 0 (totally controlled) and 6 (severely uncontrolled).
Change from baseline in Asthma Controlled Test (ACT) score | Baseline, week 4, week 8 and week 12
  1. Asthma Controlled Test (ACT); grouped in five domains; frequency of shortness of breath, general asthma symptoms, use of rescue medications, the effect of asthma on daily functioning, and overall self-assessment of asthma control. 5-point scale (for symptoms and activities: 1=all the time to 5= not at all; for asthma control rating: 1=not controlled at all to 5=completely controlled). The scores range from 5 (poor control of asthma) to 25 (complete control of asthma), with higher scores reflecting greater asthma control. An ACT score >19 indicates well-controlled asthma

SECONDARY OUTCOMES:
Change from baseline in Peak expiratory flow (PEF) | Baseline, week 4, week 8 and week 12
  The mean value of PEF (Litre per minute) for baseline, week 4, 8 and 12 was analysed.
Change from baseline in Forced Expiratory Volume in One Second (FEV1) | Baseline and week 12
  The mean value for baseline and week 12 was analysed.
Percentage of participants who were categorized from asthma controlled assessment following GINA guideline | Baseline, week 4, week 8 and week 12

CONTACTS AND LOCATIONS:
Overall Officials: Narongwit Nakwan, M.D., Study Chair — HatYai Hospital
Locations (1):
- Narongwit Nakwan, Hat Yai, Changwat Songkhla, Thailand

IPD SHARING:
Plan to Share IPD: Undecided